CLINICAL TRIAL: NCT06478160
Title: Effectiveness of Closed-blood Sampling Devices in the Adult Critically Ill Patient: Multicenter Randomized Clinical Trial
Brief Title: Closed-blood Sampling Devices in the Adult Critically Ill Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other); Hospital Universitario Rey Juan Carlos (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Virgen Macarena (Other)
Responsible Party: Principal Investigator, Marta Raurell-Torreda, Clinical Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Closed-blood sampling devices
Record Dates: First submitted 2024-06-14; First posted 2024-06-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acceptability of Health Care
Keywords: anaemia; transfusion; diagnostic blood loss; phlebotomy; blood management; hospital-acquired anemia; iatrogenic anemia; sampling practices; blood conservation; blood sample collection; catheter-related infections; critical care; nursing; blood conservation devices; clinical trial; laboratory testing; blood chemistry tests
MeSH Terms: conditions — Patient Acceptance of Health Care; Anemia; Catheter-Related Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes Assessor and statistician who analyze the results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CBSD-experimental group (Experimental): blood collection with Closed-Blood Sampling System (CBSD)
  Interventions: Device: Closed-Blood Sampling Devices
- Waste discard volume, control group (Active Comparator): Blood collection without CBSD, usual practice, need to waste discard volume
  Interventions: Other: Waste discard volume

INTERVENTIONS:
Device: Closed-Blood Sampling Devices — blood collection with Closed-Blood Sampling System (CBSD)
  Arms: CBSD-experimental group
Other: Waste discard volume — Blood collection without CBSD, usual practice, need to waste discard volume
  Arms: Waste discard volume, control group

SUMMARY:
Based on the hypothesis that the strategy of using Closed-Blood Sampling Devices (CSBD, experimental group) compared to the usual practice (waste discard volume, control group), in critically ill adult patients, will decrease the amount of blood withdrawn for laboratory tests, we want to analyze the number of red blood cells (RBC) administered and arterial catheter-related adverse events (catheter-related bacteremia, catheter obstruction, CBSD malfunction, loss of arterial pressure waveform on the patient's bedside monitor) in both study groups, during ICU stay and up to a maximum of 21 days.

DETAILED DESCRIPTION:
When a patient with an arterial catheter completes 24h of admission to the unit, with an expected catheter stay of more than 72 hours, inclusion in the study will be assessed. If the patient does not meet the non-inclusion or exclusion criteria and consents to participate in the study, he/she will be randomized to the CBSD-experimental group or waste discard volume- control group.

If the patient belongs to the CBSD-experimental group, the CBSD will be placed in the arterial line at that moment. All extractions performed will be through the arterial catheter and using the CBSD.

In the waste discard volume- control group, the arterial catheter will also be used for extractions but with the usual open extraction system of the ICU. To quantify the blood loss related to blood collection for laboratory tests, the volume of discharge (VD) used for each analysis through the arterial catheter will be recorded. In the CBSD-experimental group the VD for arterial catheter will be zero since CBSD will always be used. The laboratory tubes extracted in each analysis will also be recorded.

Data on blood analysis, blood transfusion and adverse events related to the arterial catheter will be recorded daily during the ICU stay, up to day 21 maximum and/or day of ICU discharge and/or exitus.

Patients discharged from ICU to hospitalization will be followed only during the first 48h to know if they have received red blood cell concentrates and with what previous Hemoglobine (Hb) and hematocrit (Hto).

Catheter insertion and maintenance will be carried out in the same way in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an arterial catheter who agree to participate in the study, with a stay in the ICU of 24h and a minimum of 72h more with an arterial catheter

Non-inclusion criteria: Therapeutic Limitation of Life Support, Jehovah's Witnesses.

Exclusion Criteria:

* Patients with chronic renal failure
* Patients with active gastrointestinal bleeding
* Patients diagnosed with hematologic cancer
* Women with menstruation at the time of admission
* Pregnant women

Withdrawal criteria: presence of active gastrointestinal bleeding during the study inclusion period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-06-07 (Estimated); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Units of red blood cells transfusion | Every day during the ICU stay and up to a maximum of 21 days after randomization (day 0)
  Number of red blood cells (RBC) units administered in both study groups

SECONDARY OUTCOMES:
Volume of blood drawn | Every day during ICU stay and up to a maximum of 21 days after randomization (day 0).
  Volume of blood drawn in mL for laboratory testing in both study groups
Levels of hemoglobine and hematocrit | Every day during ICU stay and up to a maximum of 21 days after randomization (day 0).
  Hemoglobin (Hb) in g/dL and hematocrit (%) in both study groups
Number and type of adverse events | Every day during the stay and up to a maximum of 21 days after randomization (day 0):
  Arterial catheter-related adverse events in both groups (infection and/or catheter obstruction; lose of arterial pressure monitoring)

CONTACTS AND LOCATIONS:
Overall Officials: Raurell-Torreda Marta, Principal Investigator — University of Barcelona
Locations (3):
- Spain (3):
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Rey Juan Carlos, Madrid, Madrid
  - Hospital Virgen de la Macarena, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vlaar AP, Oczkowski S, de Bruin S, Wijnberge M, Antonelli M, Aubron C, Aries P, Duranteau J, Juffermans NP, Meier J, Murphy GJ, Abbasciano R, Muller M, Shah A, Perner A, Rygaard S, Walsh TS, Guyatt G, Dionne JC, Cecconi M. Transfusion strategies in non-bleeding critically ill adults: a clinical practice guideline from the European Society of Intensive Care Medicine. Intensive Care Med. 2020 Apr;46(4):673-696. doi: 10.1007/s00134-019-05884-8. Epub 2020 Jan 7. PMID 31912207
- [Result] Raurell-Torreda M, Fernandez-Castillo RJ, Rodriguez-Delgado ME, Arias-Rivera S, Basco-Prado L. Best practices for iatrogenic anaemia prevention in the intensive care unit: Blood-sparing techniques. Nurs Crit Care. 2025 Jan;30(1):47-52. doi: 10.1111/nicc.13084. Epub 2024 Apr 23. PMID 38654607
- [Derived] Raurell-Torreda M, Arias-Rivera S, Fernandez-Castillo RJ, Frade-Mera MJ, Gonzalez-Caro MD, Zaragoza-Garcia I, Andreu-Vazquez C, Muriel-Garcia A; Grupo Ahorro-Sangre (Blood-Sparing Research Group). Effectiveness of Closed Blood-Sampling Devices in Critically Ill Adults: A Feasibility Trial. Nurs Crit Care. 2026 Jan;31(1):e70343. doi: 10.1111/nicc.70343. PMID 41546433